CLINICAL TRIAL: NCT04018105
Title: Influence of Preprandial Metformin Administration on Carbohydrate Absorption: Pilot Randomized Controlled Study
Brief Title: Influence of Preprandial Metformin Administration on Carbohydrate Absorption
Acronym: METTIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_35; 2019-001175-36 (EudraCT Number)
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Impaired Glucose Tolerance; Type2 Diabetes
Keywords: Impaired glucose tolerance; type 2 diabetes; obesity; carbohydrate absorption; metformin
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taking metformin 30 or 60 minutes before the OGTT (Experimental)
  Interventions: Other: Oral glucose tolerance test (OGTT) with or without metformin
- No metformin before OGTT (Placebo Comparator)
  Interventions: Other: Oral glucose tolerance test (OGTT) with or without metformin

INTERVENTIONS:
Other: Oral glucose tolerance test (OGTT) with or without metformin — Each participant will have 3 OGTT, one without metformin, one with metformin30 minutes before the test, one with metformin 60 minutes before the test. The order for each test will be randomized.

SUMMARY:
Type 2 diabetes is spreading worldwide as well as obesity. Metformin is the most prescribed antidiabetic medication. One suggested mechanism of action is by decreasing carbohydrate absorption.

It is usually recommended to take metformin during the meal to decrease gastrointestinal side effects. However, if metformin decreases carbohydrate absorption, this might not be the most efficient intake.

To study the influence of preprandial metformin administration on carbohydrate absorption, it will repeat 3 oral glucose tolerance test on obese dysglycemic patients, without metformin or with metformin administer 30 or 60 minutes before. We will also evaluate how it impacts gastrointestinal tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI ≥30 kg/m2)
* Dysglycemia (HbA1c≥ 6,0 %)
* No anti diabetic medication

Exclusion Criteria:

* No obesity (BMI < 30 kg/m2)
* No dysglycemia (HbA1c <6,0%)
* Treatment that might interfere with carbohydrate absorption (anti diabetic medication, antibiotics, probiotics, steroids)
* Anemia (Hb <12 g/dL)
* Organ failure
* Inflammatory Bowel Disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of D-Xylose | During the 3 hours OGTT

SECONDARY OUTCOMES:
Number of Participants with gastrointestinal side effects | During the 3 hours OGTT
Area under the curve of blood glucose | During the 3 hours OGTT
Area under the curve of insulin | During the 3 hours OGTT
Area under the curve of GLP-1 | During the 3 hours OGTT

CONTACTS AND LOCATIONS:
Overall Officials: camille Marciniak, MD, Principal Investigator — University Hospital, Lille